CLINICAL TRIAL: NCT04173689
Title: The Effect of Inspiratory Muscle Training and Breathing Exercises Combined With Upper Extremity and Trunk in Patients With Sarcoidosis
Acronym: physio
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Esma Yildiz, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pulmonary Sarcoidosis
Record Dates: First submitted 2019-11-07; First posted 2019-11-22 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Pulmonary Sarcoidosis
Keywords: Sarcoidosis
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratuar muscle training group (Active Comparator): This group will be given inspiratory muscle training (IMT) at home for 15 minutes twice a day for 7 days a week with the resh Threshold IMT 'device. In the IMT group, the initial training intensity will be determined by measuring the maximal inspiratory muscle strength (MRP) with the intraoral pressure measuring device, 30% of the measured MRP value will be started at the first evaluation and the new training intensity will be determined by calculating 30% of the measured value by repeating the MRP measurement every week.
  Interventions: Device: Threshold IMT
- Exercise group (Active Comparator): This group will perform upper extremity and trunk exercises combined with breathing exercises at home for 7 days, twice a day for 15 minutes. Patients in both groups will perform a single 15-minute session once a week at the hospital under the supervision of a physiotherapist.
  Interventions: Other: breathing exercises combined with upper extremity and trunk

INTERVENTIONS:
Device: Threshold IMT — 7 days a week, 2 times a day 15 min each
  Other Names: Philips
  Arms: Inspiratuar muscle training group
Other: breathing exercises combined with upper extremity and trunk — upper extremity and trunk exercises combined with breathing exercises for 7 days a week, 2 times a day for 15 minutes each
  Arms: Exercise group

SUMMARY:
This is an educational work. Thirty patients with pulmonary sarcoidosis will be included in the study and randomly selected into two training groups.One group will receive home inspiratory muscle training (IMT) for 15 minutes, twice a day, 7 days a week with the resh Threshold IMT 'device. In the IMT group, the initial training intensity will be determined by measuring the maximal inspiratory muscle strength (MIP) with the intraoral pressure measuring device, 30% of the measured (MIP) value will be started at the first evaluation and the new training intensity will be determined by calculating 30% of the measured value by repeating the MIP measurement every week. The other group will perform upper extremity and trunk exercises combined with respiratory exercises at home for 7 days, twice a day for 15 minutes.Patients will be evaluated before the training program and 8 weeks after the training. In the first evaluation, demographic information and clinical characteristics of the patients will be noted.In this study, upper and lower extremity exercise capacity, respiratory functions, peripheral muscle strength, dyspnea, fatigue, sleep quality, cognitive function, daily living activities, physical activity level, anxiety, depression, upper extremity and trunk exercises combined with inspiratory muscle training in patients with sarcoidosis and the impact on quality of life.

DETAILED DESCRIPTION:
Patients who are in stage II-III with sarcoidosis diagnosed pulmonary involvement who are admitted to the Department of Chest Diseases of Cerrahpaşa Medical Faculty Hospital of Istanbul University will be included in the 30-70 age group 6 months after systemic treatment or no treatment. Patients with stages I and IV, malignancy, heart failure, orthopedic problems and who have to undergo systemic sarcoidosis treatment during the study will not be included in the study. Thirty-four patients who meet the inclusion criteria will be included in the study by signing the informed consent form. In the first evaluation, demographic information and clinical characteristics of the patients will be noted. Lower and upper extremity functional capacities of the patients before and after training will be evaluated with 6-minute walk test (6MWT), 6-minute step test (6DST), 6-minute pegboard ring test (6DPBRT) and 30-second sit-down test. Percentage values of FVC, FEV1, FEV1 / FVC, PEF, FEF (25-75%) parameters according to measured and expected values will be recorded by performing pulmonary function test. Respiratory muscle strength will be determined by measuring maximal inspiratory pressure (MRP) and maximal expiratory pressure (MEP) with the intraoral pressure gauge. Dyspnea sensation Modified Borg and Modified Medical Research Council (MMRC) scale, fatigue state Fatigue Severity Scale (FSS), peripheral muscle strength hand dynamometer, quality of life George Respiratory Diseases Questionnaire (SGRQ), anxiety and depression status Hospital Anxiety and Depression Scale (HAD), physical activity level International Physical Activity Questionnaire-Short form (IPAQ-S), cognitive function Montreal Cognitive Assessment Scale (MOCA), daily living activities London Chest Daily Living Activities Scale and sleep quality will be evaluated with Epworth Sleepiness Scale (ESS).

ELIGIBILITY:
Inclusion Criteria:

* The study was conducted in Istanbul University Cerrahpaşa Medical Faculty Hospital Pulmonary Diseases Department with sarcoidosis diagnosed with pulmonary involvement in stage II-III,
* 6 months after receiving systemic treatment or no treatment.

Exclusion Criteria:

* Patients with stage I and IV,
* malignancy,
* heart failure,
* orthopedic problems
* who had to undergo systemic sarcoidosis treatment during the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Fatigue severity scale | 8 week
  0-7. high score shows deterioration. <2,8 no fatigue. >6,1 chronic fatigue syndrome
6 minute walk test | 8 week
  Increased walking distance in 6 minutes
Medical Research Council Dyspnea Scale | 8 week
  0-4. high score shows deterioration
Respiratory assesment | 8 week
  measure respiratory muscle strength
Epworth sleepiness scale | 8 week
  0-30. high score shows deterioration
Hospital Anxiety Scale | 8 week
  anxiety 0-21 .high score shows deterioration
Hospital Depression Scale | 8 week
  depression 0-21. high score shows deterioration
Montreal Cognitive Assessment Scale | 8 week
  assess cognitive functions of individuals.0-30. high score indicates improvement
London Chest Daily Living Activities Scale | 8 week
  Measuring daily living activities. high score shows deterioration. 0-75

CONTACTS AND LOCATIONS:
Overall Officials: Rengin DEMİR, Study Director — counselor
Locations (1):
- Esma Yıldız, Edirne, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No